CLINICAL TRIAL: NCT02569749
Title: Sleep Apnea-Hypopnea Syndrome Screening
Brief Title: Sleep Apnea Screening
Status: Terminated | Type: Observational
Why Stopped: Administrative reasons
Sponsor: Arrhythmia Network Technology S.L. (Other)
Responsible Party: Sponsor
Other Study IDs: SAHS2
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Sleep Apnea/Hypopnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: Patients with pacemaker indication (pacemaker already implanted or to be implanted)
  Interventions: Other: Berlin and Epworth questionaries; Other: Sleep apnea monitoring in those patients in whom a pacemaker with monitoring apnea system has been implanted.; Other: Night polygraph / Polysomnography
- Group 2: Patients with ICD or CRTD therapy indication (device already implanted or to be implanted)
  Interventions: Other: Berlin and Epworth questionaries; Other: Night polygraph / Polysomnography
- Group 3: Patients with heart failure an preserved LVEF (40-50%)
  Interventions: Other: Berlin and Epworth questionaries; Other: Night polygraph / Polysomnography
- Group 4: Patients with heart failure and reduced LVEF (<40%)
  Interventions: Other: Berlin and Epworth questionaries; Other: Night polygraph / Polysomnography

INTERVENTIONS:
Other: Berlin and Epworth questionaries
Other: Sleep apnea monitoring in those patients in whom a pacemaker with monitoring apnea system has been implanted.
  Groups: Group 1
Other: Night polygraph / Polysomnography

SUMMARY:
To assess the incidence of Sleep Apnea-Hypopnea Syndrome (SAHS), both obstructive and central, in patients with: 1) pacemaker indication; 2) implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRTD), 3) heart failure and preserved left ventricular ejection fraction (LVEF) and 4) heart failure and reduced LVEF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* No previous diagnosis of sleep apnea
* Fulfilling at least one of the following:

  1. Pacemaker indication
  2. ICD or CRTD therapy indication
  3. Heart failure and preserved LVEF (40-50%)
  4. Heart failure and reduced LVEF (<40%)
* Signed informed consent

Exclusion Criteria:

* Age younger than 18 years
* Renal hemodialysis
* Cardiac transplant indication
* Women who are pregnant
* Advanced cancer
* Enrollment in another investigational study
* Able and willing to comply with all testing and requirements
* Patient not suitable for inclusion due to psychiatric conditions or short life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to be included in the registry:
  * 200 patients with pacemaker indication in whom a pacemaker with sleep apnea monitoring system has been implanted.
  * 100 patients with pacemaker indication in whom a pacemaker with no sleep apnea monitoring system has been implanted.
  * 100 patients with ICD or CRDT therapy indication.
  * 100 patients with heart failure and preserved LVEF (40-50%).
  * 100 patients with heart failure and reduced LVEF (<40%).
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with SAHS in patients with pacemaker indication | 1 month
Percentage of patients with SAHS in patients with ICD or CRTD therapy | 1 month
Percentage of patients with SAHS in patients with heart failure and preserved LVEF | 1 month
Percentage of patients with SAHS in patients with reduced LVEF | 1 month

SECONDARY OUTCOMES:
Percentage of patients with obstructive sleep apnea in all groups | 1 month
Percentage of patients with central sleep apnea in all groups | 1 month

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - HM Hospitales, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid

REFERENCES:
- [Background] Young T, Evans L, Finn L, Palta M. Estimation of the clinically diagnosed proportion of sleep apnea syndrome in middle-aged men and women. Sleep. 1997 Sep;20(9):705-6. doi: 10.1093/sleep/20.9.705. PMID 9406321
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Marshall NS, Wong KK, Liu PY, Cullen SR, Knuiman MW, Grunstein RR. Sleep apnea as an independent risk factor for all-cause mortality: the Busselton Health Study. Sleep. 2008 Aug;31(8):1079-85. PMID 18714779
- [Background] Young T, Finn L, Peppard PE, Szklo-Coxe M, Austin D, Nieto FJ, Stubbs R, Hla KM. Sleep disordered breathing and mortality: eighteen-year follow-up of the Wisconsin sleep cohort. Sleep. 2008 Aug;31(8):1071-8. PMID 18714778
- [Background] Ronald J, Delaive K, Roos L, Manfreda J, Bahammam A, Kryger MH. Health care utilization in the 10 years prior to diagnosis in obstructive sleep apnea syndrome patients. Sleep. 1999 Mar 15;22(2):225-9. doi: 10.1093/sleep/22.2.225. PMID 10201067
- [Background] Fietze I, Rottig J, Quispe-Bravo S, Riedel F, Witte J, Baumann G, Witt C. Sleep apnea syndrome in patients with cardiac pacemaker. Respiration. 2000;67(3):268-71. doi: 10.1159/000029509. PMID 10867594
- [Background] Garrigue S, Pepin JL, Defaye P, Murgatroyd F, Poezevara Y, Clementy J, Levy P. High prevalence of sleep apnea syndrome in patients with long-term pacing: the European Multicenter Polysomnographic Study. Circulation. 2007 Apr 3;115(13):1703-9. doi: 10.1161/CIRCULATIONAHA.106.659706. Epub 2007 Mar 12. PMID 17353437
- [Background] Pepin JL, Chouri-Pontarollo N, Tamisier R, Levy P. Cheyne-Stokes respiration with central sleep apnoea in chronic heart failure: proposals for a diagnostic and therapeutic strategy. Sleep Med Rev. 2006 Feb;10(1):33-47. doi: 10.1016/j.smrv.2005.10.003. Epub 2005 Dec 22. PMID 16376589
- [Background] Javaheri S. Sleep disorders in systolic heart failure: a prospective study of 100 male patients. The final report. Int J Cardiol. 2006 Jan 4;106(1):21-8. doi: 10.1016/j.ijcard.2004.12.068. PMID 16321661
- [Background] Tremel F, Pepin JL, Veale D, Wuyam B, Siche JP, Mallion JM, Levy P. High prevalence and persistence of sleep apnoea in patients referred for acute left ventricular failure and medically treated over 2 months. Eur Heart J. 1999 Aug;20(16):1201-9. doi: 10.1053/euhj.1999.1546. PMID 10448029
- [Background] Defaye P, de la Cruz I, Marti-Almor J, Villuendas R, Bru P, Senechal J, Tamisier R, Pepin JL. A pacemaker transthoracic impedance sensor with an advanced algorithm to identify severe sleep apnea: the DREAM European study. Heart Rhythm. 2014 May;11(5):842-8. doi: 10.1016/j.hrthm.2014.02.011. Epub 2014 Feb 19. PMID 24561163
- [Background] Javaheri S, Parker TJ, Liming JD, Corbett WS, Nishiyama H, Wexler L, Roselle GA. Sleep apnea in 81 ambulatory male patients with stable heart failure. Types and their prevalences, consequences, and presentations. Circulation. 1998 Jun 2;97(21):2154-9. doi: 10.1161/01.cir.97.21.2154. PMID 9626176
- [Background] Arias MA, Garcia-Rio F, Alonso-Fernandez A, Sanchez AM. [Sleep apnea-hypopnea syndromes and heart failure]. Rev Esp Cardiol. 2007 Apr;60(4):415-27. Spanish. PMID 17521550
- [Background] Kasai T, Bradley TD. Obstructive sleep apnea and heart failure: pathophysiologic and therapeutic implications. J Am Coll Cardiol. 2011 Jan 11;57(2):119-27. doi: 10.1016/j.jacc.2010.08.627. PMID 21211682